CLINICAL TRIAL: NCT04122755
Title: A Single Ascending Dose, Open-Label Study Evaluating the Safety, Tolerability, And Pharmacokinetics of ALA-1000 in Opioid-Dependent Individuals
Brief Title: Single Ascending Dose Study of ALA-1000
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alar Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A1-19-P01
Record Dates: First submitted 2019-10-08; First posted 2019-10-10 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort1 (Experimental): Subjects receive a single subcutaneous injection of 1-fold ALA-1000 dose (first in human dose).
  Interventions: Drug: ALA-1000
- Cohort2 (Experimental): Subjects receive a single subcutaneous injection of 2-fold ALA-1000 dose
  Interventions: Drug: ALA-1000
- Cohort3 (Experimental): Subjects receive a single subcutaneous injection of 4.7-fold ALA-1000 dose
  Interventions: Drug: ALA-1000
- Cohort4 (Experimental): Subjects receive a single subcutaneous injection of 9.4-fold ALA-1000 dose
  Interventions: Drug: ALA-1000
- Cohort5 (Experimental): Subjects receive a single subcutaneous injection of 18.8-fold ALA-1000 dose
  Interventions: Drug: ALA-1000
- Cohort6 (Experimental): Subjects receive a single subcutaneous injection of 18.8-fold ALA-1000 dose after 7 days of buprenorphine sublingual film dosing
  Interventions: Drug: ALA-1000; Drug: buprenorphine sublingual film

INTERVENTIONS:
Drug: ALA-1000 — Blood sample for PK analysis are collected before and post single injection of ALA-1000 (Day1) according to the schedule of procedures. Subjects remain in the residential phase through Day21 for safety assessment.
  Other Names: Depot Buprenorphine Formulation
Drug: buprenorphine sublingual film — ALA-1000 injection after 7 days of buprenorphine sublingual film dosing. Blood sample for PK analysis are collected before and post sublingual buprenorphine dosing on Day-1
  Arms: Cohort6

SUMMARY:
An open-label study designed to evaluate the safety, tolerability, and pharmacokinetics of ALA-1000 in opioid-dependent subjects. To characterize the PK profile of ALA-1000 in 5 single ascending dose cohorts and a sixth cohort of single ALA-1000 after receiving buprenorphine sublingual films for 7 days.

DETAILED DESCRIPTION:
The study will include opioid-dependent subjects who have been receiving stable, orally administered buprenorphine for at least 2 weeks or buprenorphine naïve subjects who will be stabilized on orally administered buprenorphine for 3 days prior to ALA-1000 administration.

All subjects will be washed off of oral buprenorphine for 7 days prior to ALA-1000 administration except Cohort 6 which will receive ALA-1000 administration after 7 days of buprenorphine sublingual film dosing.

The subsequent cohorts will be initiated after safety and PK information from the preceding cohorts is available.

The expected maximum duration of participation for each subject is 192 days approximately, consisting of up to a 7-day screening period, up to a 31-day residential phase, and up to a 154-day nonresidential period.

ELIGIBILITY:
Inclusion Criteria:

1. Competent to provide informed consent.
2. Voluntarily provide informed consent and Health Insurance Portability and Accounting Act (HIPAA) Authorization prior to any procedures or evaluations performed specifically for the sole purpose of the study.
3. Male or female between 18 to 65 years of age inclusive at the screening visit.
4. Meets DSM-5 criteria for Opioid Use Disorder (OUD) and is seeking treatment of OUD.
5. Body Mass Index (BMI) ≥ 18 and ≤ 35 kg/m2 at screening visit.
6. Female subjects of childbearing potential must agree to use a reliable method of birth control (e.g., total abstinence, condom and spermicide, intrauterine device (IUD), oral contraception which has been stable for 30 days) and at least 120 days after stopping the investigational product.
7. Agree to withdraw from opiates for at least 12 hours prior to admission to clinical unit.
8. Agree not to take any buprenorphine product (other than ALA-1000 and buprenorphine sublingual films during tolerability/induction period) during the study.

Exclusion Criteria:

1. History or presence of a significant medical disease or disorder which, in the opinion of the investigator, increases the risk of the study drug or may confound the interpretation of study measures, as confirmed by screening laboratory results.
2. Clinically significant abnormal findings on physical examination, vital signs, or Electrocardiogram (ECG). Defined as having a QTc (Fridericia) interval > 470 msec or any other clinically significant abnormalities at screening, check-in, or prior to administration of ALA-1000.
3. Pregnant or lactating.
4. History of suicidal behavior in the past 1 year or current suicidal ideation as per investigator judgement.
5. Currently meets Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for substance use disorder, moderate or severe for any substance other than opioids, caffeine, or nicotine.
6. Currently meets criteria for any unstable psychiatric disorder, including schizophrenia, schizoaffective, bipolar disorder (depression and stable bipolar disorder are not excluded if condition has been stable for at least 60 days).
7. Current diagnosis of Acquired Immune Deficiency Syndrome (AIDS) as confirmed by Western Blot and viral load laboratory results.
8. Acute active Hepatitis B or C as evidenced by positive serology and Aspartate aminotransferase (AST)/ Alanine aminotransferase (ALT) >2 upper limit of normal (ULN)
9. History of blood donation in excess of 450 mL within 30 days prior to Visit 1.
10. Received treatment with an investigational drug or device within 90 days prior to Visit 1.
11. Use of strong inhibitors or inducers of cytochrome P450 3A4 (CYP3A4) within 30 days prior to Visit 1.
12. Use of any new medication, vitamins, or supplements within 7 days prior to Visit.
13. Hypersensitivity or allergy to buprenorphine or other opioids which, in the opinion of the investigator, would compromise subject safety.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2021-05-03 (Actual); Study Completion 2021-05-03 (Actual)

PRIMARY OUTCOMES:
Incidence of AEs will be summarized by treatment overall, by severity, and by relationship to ALA-1000. Serious AEs and AEs leading to discontinuation of study drug will also be presented. | Baseline (prior to dosing) through the End of Study (Day175), or Early termination
Change of vital signs will be assessed in subjects receiving ALA-1000. | Baseline (prior to dosing) through the End of Study (Day175), or Early termination
  Vital signs including blood pressure, pulse rate, respiration rate, pulse oximetry and temperature. Systolic and diastolic blood pressure will be assessed while supine and standing. Pulse oximetry will be monitored continuously for 24 hours post injection to assess for any signs/symptoms of respiratory depression.
Chang of clinical laboratory assessments (biochemistry, hematology and urinalysis) will be assessed in subjects receiving ALA-1000. | Baseline (prior to dosing) through the End of Study (Day175), or Early termination
  Samples will be collected for laboratory tests, including hematology, serum chemistry, urinalysis, serum/urine pregnancy test (conducted for females of childbearing potential only), and urine drug screen, to assess the safety of subjects.
Change of ECG parameter of QTcF interval will be assessed in subjects receiving ALA-1000 | Baseline (prior to dosing) through the End of Study (Day175), or Early termination
A standard physical examination will be performed to monitor the safety in subjects receiving ALA-1000 | Baseline (prior to dosing) to the End of Study (Day175), or Early termination
  The examination will include assessment of skin, head, ears, eyes, nose, throat, neck, thyroid, lungs, heart, cardiovascular, abdomen, lymph nodes, and musculoskeletal system/extremities.
Injection site assessment will be conducted to monitor the safety in subjects receiving ALA-1000 | From the end of ALA-1000 injection through the End of Study (Day175), or Early termination
  Injection site assessment including pain, tenderness, induration, erythema/redness, and swelling. If an infection develops at the injection site, the subject will be withdrawn from the study.
Concomitant medications will be reviewed and documented to monitor the safety in subjects receiving ALA-1000 | Prior to dosing through the End of Study (Day175), or Early termination
  The medication name, dose, frequency, date, and indication for use must be recorded
AUC (area under the plasma concentration-time curve) for subjects receive ALA-1000 injection | Prior to ALA-1000 injection through the End of Study (Day175), or Early termination
Cmax (maximum observed plasma concentration) for subjects receive ALA-1000 injection | Prior to ALA-1000 injection through the End of Study (Day175), or Early termination
Tmax (time to maximum concentration) for subjects receive ALA-1000 injection | Prior to ALA-1000 injection through the End of Study (Day175), or Early termination
t1/2 (time to half plasma concentration) for subjects receive ALA-1000 injection | Prior to ALA-1000 injection through the End of Study (Day175), or Early termination

SECONDARY OUTCOMES:
Change of opioid withdrawal symptoms will be assessed using Clinical Opiate Withdrawal Scale (COWS) for subjects receive ALA-1000 injection | Baseline (prior to dosing) through the End of Study (Day175), or Early termination
  Opioid withdrawal symptoms will be measured using COWS scores. Score: 5- 1 2 = mild; 1 3-24 = moderate; 25-36 = moderately severe; more than 36 = severe withdrawal
Change of suicidal ideation will be assessed using Columbia-Suicide Severity Rating Scale (C-SSRS) for subjects receive ALA-1000 injection | Screening through the End of Study (Day175), or Early termination
  Suicidal ideation scores will be reported using C-SSRS. The suicidal ideation scale identifies behaviors and thoughts that are associated with an increased risk of suicidal actions in the future. Score: 5- 1 2 = mild; 1 3-24 = moderate; 25-36 = moderately severe; more than 36 = severe suicidal ideation.
Assessment of the abstinence by urine toxicology results negative for opioids in subjects received ALA-1000 injection. | Screening through the End of Study (Day175), or Early termination

CONTACTS AND LOCATIONS:
Overall Officials: Erin Tireman, Study Director — Innovative Clinical Research
Locations (1):
- Innovative Clinical Research, Miami, Florida, United States